CLINICAL TRIAL: NCT05912426
Title: A Non-randomised Feasibility Study for a Large-scale Clinical Trial (Phase II) Testing Reduced-sodium Salt for the Prevention of the Rise in Blood Pressure With Age Among Children and Adults (6+ Years) in Nigeria (RAISED)
Brief Title: Preventing the Rise in Blood Pressure With Age Using Reduced-sodium Salt
Acronym: RAISED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University of Abuja Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HC230273; UATH/HREC/PR/2023/06/084 (Other: University of Abuja Teaching Hospital HREC)
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure
Keywords: Reduced-sodium salt; Potassium-enriched salt; Salt reduction; Blood pressure; Salt; Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced-sodium potassium-enriched salt (Experimental): Reduced-sodium potassium-enriched salt
  Interventions: Behavioral: Reduced-sodium potassium-enriched salt

INTERVENTIONS:
Behavioral: Reduced-sodium potassium-enriched salt — Supply and use of a reduced-sodium, potassium-enriched iodised salt (66% potassium chloride, 34% sodium chloride).

SUMMARY:
The study is a small-scale, short-term unblinded feasibility study to explore the acceptability and feasibility of implementing a reduced-sodium iodised salt intervention in Nigeria. This study will be used to inform a large-scale intervention trial comparing the effects of reduced-sodium salt versus regular salt on the rise in blood pressure with age.

DETAILED DESCRIPTION:
Reduced-sodium salts are a proven method for reducing sodium intake and lowering blood pressure. No studies to date have tested the effects of sodium reduction on the rise in blood pressure with age during adulthood or the critical periods of childhood and adolescence. The investigators want to explore whether reducing dietary sodium intake using reduced-sodium salt in comparison to regular salt, will attenuate the rise in blood pressure with age. This feasibility study aims to determine the feasibility of implementing a reduced-sodium iodised salt (66% potassium chloride, 34% sodium chloride) intervention in Nigeria. Specifically, the investigators will explore the feasibility of recruiting households with at least one child or adolescent 6-17 years of age and one adult ≥18 years, the acceptability of the reduced-sodium salt intervention, adherence to study procedures and data collection methods, and the effect of the reduced-sodium salt intervention on blood pressure. Secondary outcomes include household eligibility, household composition, willingness to engage in monthly follow-up visits in a longer-term trial, blood pressure, urinary sodium and potassium concentrations, height and weight. This study will be used to inform a large-scale intervention trial comparing the effects of reduced-sodium salt versus regular salt on the rise in blood pressure with age. The study will be conducted in two rural communities in Nigeria and will recruit 30 households (approximately 150 participants). All participants will be provided with the reduced-sodium salt intervention to replace all regular salt used for cooking, seasoning and food preservation over a 2-month period; there will be no control. Follow-up visits will be at 1 month and 2 months after the baseline visit, conducted either at the home or a local community healthcare centre.

ELIGIBILITY:
Inclusion Criteria:

* At least one household member is a child or adolescent (6-17 years) and at least one household member is an adult (≥18 years)
* All household members consume greater than half of meals as food prepared in the home (self-report)
* All household members provide signed informed consent/assent (consent obtained from legal guardians for those <18 years of age; assent also obtained from children/adolescents ≥12 years of age)

Exclusion Criteria:

* Any household member has serious renal impairment.
* Any household member uses a potassium-sparing diuretic.
* Any household member uses a potassium supplement.
* Any household member has other reason for concern about the use of reduced-sodium salt.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | 2 months
  Measured as the number of households recruited each month
Adherence to the reduced-sodium salt intervention | 2 months
  Measured as the self-reported proportion of regular salt replaced with intervention salt at each follow-up visit. The investigators will also estimate the quantity of intervention salt used by the household at each follow-up visit by visually estimating the amount of intervention salt that remains unused.
Acceptability of the reduced-sodium salt intervention | 2 months
  Measured as the percentage of participants that identify 'good', 'really good' or 'super good' on a brief questionnaire administered at the 2-month follow-up visit
Completion rate of visits | 2 months
  Measured as the percentage of participants that provide key data points (e.g., blood pressure, safety) at each visit

SECONDARY OUTCOMES:
Total number and percentage of households eligible to participate in the study | 2 months
  Measured as the number of eligible households over the number of households approached at registration visits.
Average number of participants per household and breakdown by age group | 2 months
Willingness to engage in monthly follow-up visits in a longer-term trial (48-months) | 2 months
  Measured as the percentage of participants that identify as 'willing', 'very willing' or 'super willing' on a brief questionnaire administered at the 2-month follow-up visit
Systolic and diastolic blood pressure | 2 months
  Measured using validated and automated sphygmomanometers, according to standard practices and definitions outlined in the Global Alliance for Chronic Disease (GACD) data dictionary
Urinary sodium concentration | 2 months
  Measured as the mmol/L of sodium from a spot urine sample
Urinary potassium concentration | 2 months
  Measured as the mmol/L of potassium from a spot urine sample
Weight | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Katrina Kissock, PhD, Study Chair — The George Institute; Bruce Neal, PhD, Principal Investigator — The George Institute; Dike Ojji, PhD, Study Director — University of Abuja Teaching Hospital
Locations (2):
- Nigeria (2):
  - Gofidna, Abuja Municipal Area Council, Federal Capital Territory
  - Jahi-2, Abuja Municipal Area Council, Federal Capital Territory

IPD SHARING:
Plan to Share IPD: Yes
Data may be used for future research purposes or shared with other researchers. Researchers wishing to obtain data for secondary research purposes must place a request with the Principal Investigator (Prof Bruce Neal) and provide a copy of their ethics approval. If the request is approved, the Principal Investigator will provide remote access to the data to other researchers via a remote data access service. All data will be made available in a de-identified format with unique participant and household Identifier (ID) numbers. Data linking participant and household IDs to identifiable participant information will not be provided.

REFERENCES:
- [Derived] Kissock KR, Okoro C, Trieu K, Ripiye NR, Orji A, Huffman MD, Neal B, Ojji D. A feasibility study for a trial testing the effects of reduced-sodium salt on the rise in blood pressure with age. Nutr Metab Cardiovasc Dis. 2025 Oct;35(10):104129. doi: 10.1016/j.numecd.2025.104129. Epub 2025 May 11. PMID 40451676